CLINICAL TRIAL: NCT03743649
Title: Strategies for Persistent Agitated Delirium in Palliative Care
Brief Title: Haloperidol and Lorazepam in Controlling Symptoms of Persistent Agitated Delirium in Patients With Advanced Cancer Undergoing Palliative Care
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2018-0706; NCI-2018-02438 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0706 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-11-09; First posted 2018-11-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Delirium; Locally Advanced Malignant Neoplasm; Metastatic Malignant Neoplasm; Recurrent Malignant Neoplasm
MeSH Terms: conditions — Delirium; Neoplasm Metastasis; Recurrence | interventions — Haloperidol; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group I (haloperidol, placebo) (Experimental): Patients receive haloperidol IV over 3-15 minutes every 4 hours and then every hour as needed and placebo IV every 4 hours and then every hour as needed until discharge from palliative care unit.
  Interventions: Drug: Haloperidol; Other: Placebo; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (lorazepam, placebo) (Experimental): Patients receive lorazepam IV over 3-15 minutes every 4 hours and then every hour as needed and placebo IV every 4 hours and then every hour as needed until discharge from palliative care unit.
  Interventions: Drug: Lorazepam; Other: Placebo; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group III (haloperidol, lorazepam) (Experimental): Patients receive haloperidol IV over 3-15 minutes every 4 hours and then every hour as needed and lorazepam IV over 3-15 minutes every 4 hours and then every hour as needed until discharge from palliative care unit.
  Interventions: Drug: Haloperidol; Drug: Lorazepam; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group IV (placebo, lorazepam) (Experimental): Patients receive two different placebos IV every 4 hours. Patients then receive placebo IV and lorazepam IV over 3-15 minutes every hour as needed until discharge from palliative care unit.
  Interventions: Drug: Lorazepam; Other: Placebo; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Haloperidol — Given IV
  Other Names: Haldol; McN-JR-1625; R 1625; R-1625
  Arms: Group I (haloperidol, placebo); Group III (haloperidol, lorazepam)
Drug: Lorazepam — Given IV
  Other Names: Ativan
  Arms: Group II (lorazepam, placebo); Group III (haloperidol, lorazepam); Group IV (placebo, lorazepam)
Other: Placebo — Given IV
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Group I (haloperidol, placebo); Group II (lorazepam, placebo); Group IV (placebo, lorazepam)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II/IIII trial studies how well haloperidol and lorazepam work in controlling symptoms of persistent agitated delirium in patients with cancer that has spread to other places in the body undergoing palliative care. Haloperidol and lorazepam may help in controlling symptoms of agitated delirium in patients with cancer and may lessen any distress that their caregivers may be experiencing.

DETAILED DESCRIPTION:
Primary Objectives:

I. To compare the effect of neuroleptic dose escalation, benzodiazepine rotation, combination therapy, and neuroleptic withdrawal on the change in the Richmond Agitation Sedation Scale (RASS) score over 24 hours in patients admitted to an acute palliative care unit (APCU) who do not respond to low-dose haloperidol

Secondary Objectives:

I. To compare the effects of neuroleptic dose escalation, benzodiazepine rotation, combination therapy, and neuroleptic withdrawal on (1) rescue medication use; (2) the proportion of patients in the target RASS range (defined as RASS between -2 and 0) as well as the proportion of patients achieving treatment response (defined as RASS reduction of ≥ 1.5 points); (3) perceived comfort as assessed by caregivers and bedside nurses; (4) delirium-related distress in caregivers and nurses (Delirium Experience Questionnaire); (5) achievement of the proxy comfort goal; (6) symptom expression (Edmonton Symptom Assessment Scale [ESAS]); (7) delirium severity (Memorial Delirium Assessment Scale [MDAS]); (8) adverse effects; and (9) quality of end-of-life care.

II. To identify novel predictive markers of response to haloperidol and lorazepam.

OUTLINE: Patients are randomized to 1 of 4 groups.

GROUP I: Patients receive haloperidol intravenously (IV) over 3-15 minutes every 4 hours and then every hour as needed and placebo IV every 4 hours and then every hour as needed until discharge from palliative care unit.

GROUP II: Patients receive lorazepam IV over 3-15 minutes every 4 hours and then every hour as needed and placebo IV every 4 hours and then every hour as needed until discharge from palliative care unit.

GROUP III: Patients receive haloperidol IV over 3-15 minutes every 4 hours and then every hour as needed and lorazepam IV over 3-15 minutes every 4 hours and then every hour as needed until discharge from palliative care unit.

GROUP IV: Patients receive two different placebos IV every 4 hours. Patients then receive placebo IV and lorazepam IV over 3-15 minutes every hour as needed until discharge from palliative care unit.

ELIGIBILITY:
Inclusion Criteria:

1. [Patients] Diagnosis of advanced cancer (defined as locally advanced, metastatic recurrent, or incurable disease)
2. [Patients] Admitted to the acute palliative care unit‡
3. [Patients] Delirium as per DSM-5 criteria
4. [Patients] Hyperactive or mixed delirium with RASS ≥1* in the past 24 h despite efforts to treat potential underlying causes
5. [Patients] On scheduled haloperidol for delirium (≤8 mg in the past 24 h) or required ≥4 mg of rescue haloperidol for agitation in the past 24 h
6. [Patients] Age 18 years or older
7. [Caregivers] Patient's spouse, adult child, sibling, parent, other relative, or significant other (partner as defined by patient)
8. [Caregivers] Age 18 years or older

Exclusion Criteria:

1. [Patients] History of myasthenia gravis or acute narrow angle glaucoma
2. [Patients] History of neuroleptic malignant syndrome or active seizure disorder (with seizure episode within the past week)
3. [Patients] History of Parkinson's disease, Alzheimer's or Lewy body dementia
4. [Patients] History of prolonged QTc or QTcF interval (>500 ms)† if documented by most recent ECG within the past month
5. [Patients] History of hypersensitivity to haloperidol or lorazepam
6. [Patients] On scheduled lorazepam within the past 48 h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Richmond Agitation Sedation Scale (RASS) score in patients admitted to an acute palliative care unit (APCU) | Baseline to 24 hours
  The effect of neuroleptic dose escalation, benzodiazepine rotation, combination therapy, and neuroleptic withdrawal will be compared on the change in the RASS score over 24 hours in patients admitted to an APCU who do not respond to low-dose haloperidol.(RASS between -2 and 0) Will use 2-sided t-tests for four pre-specified paired comparisons, if the required assumptions for this model are met. Non-parametric methods such as Wilcoxon rank-sum test may be used if any assumptions are violated.

SECONDARY OUTCOMES:
Rescue medication use | At 24 hours
  Will conduct Bonferroni adjustment for the number of rescue doses. Will perform a comparison among the four arms using analysis of variance (ANOVA), followed by selected pairwise t-test comparisons, or the Kruskal-Wallis test followed by pairwise Wilcoxon rank-sum tests if the data violate assumptions for ANOVA. Will also compare these outcomes longitudinally using linear mixed models, with treatment as a between-patient factor and time as a within-subject factor. Appropriate transformations will be used as needed to satisfy model assumptions.
Proportion of patients in the target RASS range (defined as RASS between -2 and 0) as well as the proportion of patients achieving treatment response (defined as RASS reduction of >= 1.5 points) | At 24 hours
  Will compare the proportions across all four treatment groups using a chi-squared test, followed by selected pairwise chi-squared tests. We will also compare these outcomes longitudinally and include all data after treatment administration using generalized linear mixed models, with treatment as a between-patient factor and time as a within-subject factor.
Perceived comfort as assessed by caregivers and bedside nurses questionnaire | At 24 hours
  Will be used for patients with caregivers or nurses listing "agree" or "strongly agree" for patient comfort, proportion of patients with at least 2 on the Udvalg for Kliniske Undersogelser (UKU) scale, and proportion of patients with caregivers listing "excellent" quality of end-of-life care)
Delirium-related distress in caregivers and nurses assessed using Delirium Experience Questionnaire | At 24 hours
  Examines both the recalled frequency of 6 delirium symptoms and associated distress in the rater: disorientation to time and place, visual/tactile/auditory hallucinations, delusional thoughts, and psychomotor agitation. It will be administered to family caregivers and nurses daily. The score for recalled frequency ranges between 0 and 4, where 0=not present, 1=a little of the time, 2=some of the time, 3=good part of the time, and 4=most or all of the time. The score for distress in the rater related to each delirium symptom also ranges from 0 to 4, where 0=no distress, 1=a little, 2=a fair amount, 3=very much, and 4=extremely distressed. This assessment will be administered to the blinded caregivers and bedside nurses daily.
Proxy comfort goal level | Up to 24 hours
  The achievement of the proxy comfort goal will be assessed.
Symptom expression assessed using Edmonton Symptom Assessment Scale | At 24 hours
  Validated and widely used in different clinical settings, including the APCU. It assesses the average symptom intensity of 10 symptoms (pain, fatigue, nausea, depression, anxiety, drowsiness, shortness of breath, appetite, sleep, and feeling of well-being) over the past 24 hours using an 11-point numeric rating scale, ranging from 0 (none) to 10 (worst). Because all patients will be delirious, caregivers will be asked to provide their proxy rating of ESAS daily.
Delirium severity assessed using Memorial Delirium Assessment Scale | At 24 hours
  Will perform a comparison among the four arms using ANOVA, followed by selected pairwise t-test comparisons, or the Kruskal-Wallis test followed by pairwise Wilcoxon rank-sum tests if the data violate assumptions for ANOVA. Will also compare these outcomes longitudinally using linear mixed models, with treatment as a between-patient factor and time as a within-subject factor. Appropriate transformations will be used as needed to satisfy model assumptions.
Incidence of adverse events | Up to 24 hours
Quality of end-of-life care: questionnaire | 4-8 weeks
  Will phone the bereaved caregivers who were most involved in the patient's care within 4-8 weeks of the patient's death to assess the patient's perceived quality of care and quality of life at the end-of-life, on the basis of questions previously used in the Coping with Cancer Study. Specifically, will ask caregivers, "Overall, how would you rate the care (the patient) received at the palliative care unit? Would you say it was excellent, very good, good, fair, or poor?" and "In your opinion, how would you rate the overall quality of (the patient)'s death or last week of life?" using a numeric rating scale from 0 (worst possible) to 10 (best possible). Will also ask them 2 questions related to control of agitation, adapted from the Quality of Death and Dying Questionnaire.
To identify novel predictive markers of response to haloperidol and lorazepam. | Up to 24 hours
  In each of the groups, will identify independent factors that are predictive of response (i.e. RASS reduction of >= 1.5 points) to treatment using multivariable logistic regression analysis. Will assess the predictive value of plasma biomarkers (i.e. IL-6, IL-8, IL-10, and S100B) in the subset of patients.

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (2):
  - M D Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
- Hosptial de Cancer de Barretos, Barretos, São Paulo, Brazil

REFERENCES:
- [Derived] Hui D, De La Rosa A, Tsai JS, Cheng SY, Del Fabbro E, Thomas Kuzhiyil AT, Rowe K, Azhar A, Nguyen T, Tang M, Yao CA, Huang HL, Peng JK, Hu WY, Admane S, Dev R, Chen M, Bramati P, Shete S, Bruera E. Proportional Sedation for Persistent Agitated Delirium in Palliative Care: A Randomized Clinical Trial. JAMA Oncol. 2025 Sep 1;11(9):1031-1043. doi: 10.1001/jamaoncol.2025.2212. PMID 40742738
- See also: MD Anderson Cancer Center — http://www.mdanderson.org